CLINICAL TRIAL: NCT01225380
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating 16 and 24 Weeks of Response Guided Therapy With GS-9190, GS-9256, Ribavirin (Copegus®) and Peginterferon Alfa 2a (Pegasys®) in Treatment Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection (Protocol No. GS-US-196-0123)
Brief Title: A Study of Response-Guided Duration of Combination Therapy With GS-9190, GS-9256, Pegasys® and Copegus® in Previously Untreated Subjects With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-196-0123
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; HCV RNA; Polymerase inhibitor; Protease inhibitor; Treatment naïve; GS-9190; GS-9256
MeSH Terms: conditions — Hepatitis C | interventions — tegobuvir; GS-9256; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): GS-9190 and GS-9256 in combination with Pegasys® and Copegus® for 16 or 24 weeks; Pegasys® and Copegus® may be continued for up to 48 weeks total duration depending on individual response to therapy
  Interventions: Drug: GS-9190; Drug: GS-9256; Biological: Pegasys®; Drug: Copegus®
- Arm 2 (Experimental): GS-9256 (active) and placebo matching GS-9190 in combination with Pegasys® and Copegus® for 24 weeks; Pegasys® and Copegus® may be continued for up to 48 weeks total duration depending on individual response to therapy
  Interventions: Drug: GS-9190 placebo; Drug: GS-9256; Biological: Pegasys®; Drug: Copegus®
- Arm 3 (Placebo Comparator): Placebo matching GS-9190 and placebo matching GS-9256 in combination with Pegasys® and Copegus® for 24 weeks; Pegasys® and Copegus® will be continued for up to 48 weeks total duration
  Interventions: Drug: GS-9190 placebo; Drug: GS-9256 placebo; Biological: Pegasys®; Drug: Copegus®

INTERVENTIONS:
Drug: GS-9190 — GS-9190 capsule, 20 mg BID, 16 or 24 weeks
  Arms: Arm 1
Drug: GS-9256 — GS-9256 capsule, 150 mg BID, 16 or 24 weeks
  Arms: Arm 1
Biological: Pegasys® — peginterferon alfa-2a, (solution for injection) 180 µg/week, up to 48 weeks
  Arms: Arm 1
Drug: Copegus® — ribavirin 200 mg tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day >/= 75 kg) divided twice daily (BID), up to 48 weeks
  Arms: Arm 1
Drug: GS-9190 placebo — placebo matching GS-9190 capsule BID, 24 weeks
  Arms: Arm 2
Drug: GS-9256 — GS-9256 capsule, 150 mg BID, 24 weeks
  Arms: Arm 2
Biological: Pegasys® — peginterferon alfa-2a (solution for injection) 180 µg/week, up to 48 weeks
  Arms: Arm 2
Drug: Copegus® — ribavirin 200 mg tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day >/= 75 kg) divided twice daily (BID), up to 48 weeks
  Arms: Arm 2
Drug: GS-9190 placebo — placebo matching GS-9190 capsule BID, 24 weeks
  Arms: Arm 3
Drug: GS-9256 placebo — placebo matching GS-9256 capsule BID, 24 weeks
  Arms: Arm 3
Biological: Pegasys® — peginterferon alfa-2a (solution for injection) 180 µg/week, 48 weeks
  Arms: Arm 3
Drug: Copegus® — ribavirin 200 mg tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day >/= 75 kg) divided twice daily (BID), 48 weeks
  Arms: Arm 3

SUMMARY:
This phase 2b study will evaluate the efficacy and safety of 16 and 24 weeks of response-guided duration of therapy with GS-9190 and GS-9256 in combination with Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®). Additionally, the efficacy and safety of 24 weeks of GS-9256 in combination with Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 to 70 years of age
* Chronic HCV infection for at least 6 months prior to Baseline (Day 1)
* Liver biopsy results (performed no more than 2 years prior to Screening) indicating the absence of cirrhosis
* Monoinfection with HCV genotype 1a or 1b
* HCV treatment-naïve
* Body mass index (BMI) between 18 and 36 kg/m2
* Creatinine clearance >/= 50 mL/min
* Subject agrees to use highly effective contraception methods if female of childbearing potential or sexually active male.
* Screening laboratory values within defined thresholds for ALT, AST, leukopenia, neutropenia, anemia, thrombocytopenia, thyroid stimulating hormone (TSH), potassium, magnesium

Exclusion Criteria:

* Autoimmune disease
* Decompensated liver disease or cirrhosis
* Poorly controlled diabetes mellitus
* Severe psychiatric illness
* Severe chronic obstructive pulmonary disease (COPD)
* Serological evidence of co-infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or another HCV genotype
* Suspicion of hepatocellular carcinoma or other malignancy (with exception of certain skin cancers)
* History of hemoglobinopathy
* Known retinal disease
* Subjects who are immunosuppressed
* Subjects with known, current use of amphetamines, cocaine, opiates (i.e., morphine, heroin), methadone, or ongoing alcohol abuse
* Subjects who are on or are expected to be on a potent cytochrome P450 (CYP) 3A4 or Pgp inhibitor, or a QT prolonging medication within 2 weeks of Baseline (Day 1) or during the study
* Subjects must have no history of clinically significant cardiac disease, including a family history of Long QT syndrome, and no relevant electrocardiogram (ECG) abnormalities at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) defined as undetectable HCV RNA 24 weeks after treatment cessation | 24 weeks of off-treatment follow-up

SECONDARY OUTCOMES:
Safety and tolerability of therapy as measured by frequency of laboratory abnormalities, reported adverse events, and discontinuations due to adverse events | Through up to 48 weeks treatment period and 24 weeks of off-treatment follow-up
Emergence of viral resistance following initiation of therapy with GS-9190 and GS-9256 | Through up to 48 weeks treatment period, 24 weeks of off-treatment follow-up, and up to 48 weeks of follow-up in the Resistance Registry Substudy
Viral dynamics and steady state pharmacokinetics of GS-9190 and GS-9256 when administered in combination with PEG and RBV; measured by HCV RNA levels and plasma concentrations of GS-9190 and GS-9256 over time | Through Week 4 of therapy
Long-term assessment of plasma HCV RNA in subjects who achieve SVR | 36 months following Week 72
  Plasma HCV RNA will be measured at approximately 6, 12, 24, and 36 months after Week 72.

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, Study Director — Gilead Sciences
Locations (114):
- United States (36):
  - Mayo Clinic, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - South Denver Gastroenterology, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Bach and Godofsky Infectious Diseases, Sarasota, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Emory University, Infectious Disease Clinic, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Southwest CARE Center, Santa Fe, New Mexico
  - North Shore University Hospital, Great Neck, New York
  - Concorde Medical Group, New York, New York
  - Cornell University Gastroenterology & Hepatology, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University Gastroenterology, Providence, Rhode Island
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - The North Texas Research Institute, Arlington, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Liver Institute of Virginia, Bon Secours, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Digestive Disease Institute, Seattle, Washington
- Austria (5):
  - Medizinische Universität Graz, Graz
  - LKH Innsbruck, Innsbruck
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - AKH der Stadt Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- Belgium (5):
  - SGS - Clinical Pharmacology Unit Antwerpen, Antwerp
  - ULB Erasme, Brussels
  - UCL Saint Luc, Brussels
  - UZ Antwerp, Edegem
  - CHU Sart Tilman, Liège
- Canada (10):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Division of Gastroenterology, Edmonton, Alberta
  - Downtown ID Clinic, Vancouver, British Columbia
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - John Buhler Research Centre, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Division of Infectious Diseases, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
- Czechia (6):
  - University Hospital Brno, Brno
  - Melnik Hospital, Mělník
  - University Hospital Plzen, Pilsen
  - Klinmed, s.r.o., Prague
  - Institute of Clinic and Experimental Medicine, Prague
  - Association of Physicians for Infection Diseases, Ústí nad Labem
- France (6):
  - Beaujon Hospital, Clichy
  - Henri Mondor Hospital, Créteil
  - Claude Huriez Hospital, Lille
  - Hotel Dieu Hospital, Lyon
  - Saint Joseph Hospital, Marseille
  - Nancy University Hospital Center, Vandœuvre-lès-Nancy
- Germany (11):
  - Charite University Medicine, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt/M
  - University Hospital Freiburg, Freiburg im Breisgau
  - Ifi - Institut fuer Interdisziplinaere Medizin - Studien und Projekte GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University hospital Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - Johannes Gutenberg University Hospital, Mainz
  - Ludwig-Maximilians-University Munich, München
- Italy (6):
  - Epatologia, Azienda Ospedaliero "Spedali Civili", Brescia
  - U.O. Gastroenterologia 1 - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Medicina Generale - Azienda Ospedaliera di Padova, Padua
  - U. O. C. di Gastroenterologia - Azienda Ospedaliero-Universitaria Policlinico Paolo Giaccone, Palermo
  - Unità di Malattie Infettive ed Epatologia, Azienda Ospedaliero-Universitaria, Parma
  - Gastroepatologia - Azienda Ospedaliero-Universitaria S. Giovanni Battista, Torino
- Poland (14):
  - Wojewodzki Szpital Specjalistyczny im. K. Dluskiego Oddzial Obserwacyjno-Zakazny, Bialystok
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza Oddział Obserwacyjno-Zakazny, Bydgoszcz
  - Szpital Specjalistyczny w Chorzowie, Chorzów
  - Niepubliczny Zaklad Opieki Zdrowotnej "Pol-SaNa-Med" Spolka z ograniczona odpowiedzialnoscia, Czeladź
  - Wojewodzki Szpital Zespolony w Kielcach, Kielce
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Specjalistyczny Szpital im. Dr Wl. Bieganskiego w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Radomski Szpital Specjalistyczny im. Dr Tytusa Chalubinskiego Oddzial obserwacyjno-zakazny z odcinkiem jednego dnia leczenia chorob watroby, Radom
  - Samodzielny Publiczny Wojewodzki Szpital Zespolony w Szczecinie, Szczecin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Zakazny Oddzial Dzienny, Warsaw
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Zakazny Oddział X, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw
  - EMC Instytut Medyczny S.A., Wroclaw
- Spain (6):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínico Universitario San Cecilio, Granada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ntra. Sra. de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (9):
  - Queen Elizabeth Hospital, Birmingham
  - North Manchester General Hospital, Greater Manchester
  - Royal Liverpool University Hospital, Liverpool
  - Barts and The London Hospital, London
  - University College London Hospital, London
  - Kings College Hospital, London
  - Chelsea and Westminster Hospital, London
  - Institute of Cellular Medicine (Hepatology), Newcastle upon Tyne
  - Derriford Hospital, Plymouth